CLINICAL TRIAL: NCT03251560
Title: The Clinical Effect of Fuke Qianjin Capsule on Chronic Pelvic Pain Caused by Pelvic Inflammation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aijun Sun (Other)
Collaborators: Second Hospital of Jilin University (Other); Shenzhen maternal and child health care hospital (Unknown); Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor-Investigator, Aijun Sun, professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID201706
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Chronic Pelvic Pain
Keywords: Fuke Qianjin capsule; chronic pelvic pain

STUDY DESIGN:
Intervention Model Description: half of the participants will receive Fuke Qianjin capsule, the other half participants will receive placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuke Qianjin capsule (Experimental): Fuke Qianjin capsule, 2 pills each time,three times a day, orally (0.4g/pill）,for 2months,
  Interventions: Drug: Fuke Qianjin capsule
- Placebo oral capsule (Placebo Comparator): placebo pills, 2 pills each time,three times a day, orally, for 2months
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Fuke Qianjin capsule — Fuke Qianjin capsule 0.8g pills by mouth, three times daily
  Arms: Fuke Qianjin capsule
Drug: Placebo oral capsule — Placebo oral capsule 0.8g pill by mouth, three times daily
  Arms: Placebo oral capsule

SUMMARY:
A prospective random control clinical trials to research Fuke Qianjin capsule's effects on ameliorating the pain caused by chronic pelvic disease.

DETAILED DESCRIPTION:
Fuke Qianjin capsule has been widely used in clinical medicine to ameliorate the pain caused by chronic pelvic disease.But random control trials on its effects are few.Our study was designed as a prospective random control clinical trials to research its effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female between the age of 18 and 50.
* Subject with a history of pelvic inflammatory disease suffered from one of the symptoms below and one of the signs below: symptoms:1.lower abdominal distension or pain;2.lumbosacral soreness. signs:1. enlarged,cable strip-like fallopian tube with mild tenderness palpated on one side or both sides of the uterine;2.restricted movement or adhesion fixed of the uterine;3.the sacral ligaments thicken and harden with mild tenderness.
* Subject VAS score of pelvic pain ≥4
* Subject without fertility requirements in 2 months
* Subject provides written informed consent.

Exclusion Criteria:

* Subject underwent recurrent urinary system infection or interstitial cystitis
* Subject underwent irritable bowel syndrome
* Subject has other complications in addition to chronic pelvis inflammation diseases leading to chronic pelvic pain,such as gynecological malignant disease,irregular vaginal bleeding, endometriosis,adenomyosis,ovarian neoplasm with a diameter >5cm by ultrasound
* Subject is pregnant or lactating.
* Subject has a severe systemic disease, such as cardiovascular system
* Subject has a history of malignancy or radiotherapy.
* Subject has undergone any chronic pelvic pain treatment including antibiotics,paregoric,physiotherapy or any other related treatment within 1month prior to randomization.
* Subject has mental disorder incapable of elementary cooperations.
* Subject has an allergic history to the experimental drug.
* Subject has participated in other clinical researches of medicine within 1month prior to randomization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 240 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale Score(VAS score) of pelvic pain | 5 minutes
  pelvic pain degree related assessment
C-reaction protein(CRP) | 5 minutes
  inflammation response biomarker assessment
Interleukin 6 (IL-6) | 5 minutes
  pro-inflammatory cytokine assessment
Tumor necrosis factor alpha (TNFα) | 5 minutes
  systemic inflammation biomarker assessment

SECONDARY OUTCOMES:
The Short Form (36) Health Survey (SF-36) | 5 minutes
  health status measure
Short-form McGill Pain Questionnaire (SF-MPQ) | 5 minutes
  pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Aijun Sun, MD, Principal Investigator — Peking Union Medical College Hospital,Peking Union Medical College,Chinese Academy of Medical Sciences
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within 2 months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel.Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Steege JF, Siedhoff MT. Chronic pelvic pain. Obstet Gynecol. 2014 Sep;124(3):616-629. doi: 10.1097/AOG.0000000000000417. PMID 25162265
- See also: Causes of chronic pelvic pain in women — https://www.uptodate.com/contents/causes-of-chronic-pelvic-pain-in-women?source=Out%20of%20date%20-%20zh-Hans&search=%E6%85%A2%E6%80%A7%E7%9B%86%E8%85%94%E7%82%8E&selectedTitle=4~150
- See also: Chronic Pelvic Inflammatory Disease — https://www.clinicalkey.com/#!/content/book/3-s2.0-B9781455770083000053?scrollTo=%23hl0001217